CLINICAL TRIAL: NCT01793233
Title: Longitudinal Assessment of Ovarian Reserve in Adolescents With Lymphoma
Brief Title: Blood Sample Markers of Reproductive Hormones in Assessing Ovarian Reserve in Younger Patients With Newly Diagnosed Lymphomas
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ALTE11C1; NCI-2013-00069 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ALTE11C1 (Other: Children's Oncology Group); COG-ALTE11C1 (Other: DCP); ALTE11C1 (Other: CTEP); U10CA095861 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Anaplastic Large Cell Lymphoma; Burkitt Lymphoma; Diffuse Large B-Cell Lymphoma; Hodgkin Lymphoma; Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease; Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ancillary-Correlative (menstrual diary, biomarker analysis): Patients complete a menstrual diary to document vaginal bleeding and undergo blood sample collections at baseline, the 3rd course of chemotherapy, at the end of chemotherapy, and at 6 and 12 months post-treatment.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies blood sample markers of reproductive hormones in assessing ovarian reserve in younger patients with newly diagnosed lymphomas. Studying samples of blood from patients with cancer in the laboratory may help measure the effect of curative therapy for lymphoma on ovarian failure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare anti mullerian hormone (AMH), follicle stimulating hormone (FSH), and estradiol (E2) between patients at baseline and cross section of controls and again between patients at 12 months off therapy and cross section of controls.

II. Describe the trajectory of AMH, FSH, and E2 from baseline to 12 months after completion of gonadotoxic cancer treatment.

III. Evaluate degree of change of AMH/FSH/E2 from baseline to end of therapy in patients.

IV. Evaluate degree of recovery of AMH/FSH/E2 from end of therapy to 12 months off therapy.

SECONDARY OBJECTIVES:

I. Describe acute ovarian failure (AOF) prevalence 12 months post-therapy. II. Collect blood samples for future evaluation of drug metabolizing enzyme polymorphisms.

OUTLINE:

Patients complete a menstrual diary to document vaginal bleeding and undergo blood sample collection at baseline, the 3rd course of chemotherapy, at the end of chemotherapy, and at 6 and 12 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had first menses >= 6 months prior to enrollment
* Patients must be newly diagnosed with lymphoma; this includes but is not limited to Hodgkin lymphoma, Burkitts lymphoma, diffuse large B cell lymphoma, and anaplastic large cell lymphoma
* Planned cancer treatment must include an alkylating agent: i.e. procarbazine, cyclophosphamide, ifosphamide; planned cancer treatment must be less than one year
* Patients with any performance status are eligible for enrollment
* Patients may take hormone medications excluding gonadotropin-releasing hormone (GnRH) analogues
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients who have previously received chemotherapy other than steroids and intrathecal chemotherapy are not eligible
* Patients who have a secondary malignancy are not eligible
* Patients with known history of ovarian disease: e.g. Turner syndrome or polycystic ovarian syndrome are not eligible
* Patients in whom planned therapy includes: removal or uterus or ovary(ies), pelvic irradiation, cranial irradiation or hematopoietic stem cell transplantation are not eligible
* Patients who previously have had their uterus or ovary(ies) removed are not eligible
* Patients who have received gonadotropin release hormone agonist or antagonist (e.g. Lupron) prior to study entry are not eligible
* Patients who are pregnant or breast feeding are not eligible
* Patients who have undergone or are planning to undergo ovarian tissue, oocyte or embryo cryopreservation prior to treatment are not eligible

Max Age: 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with newly diagnosed lymphoma at Children's Oncology Group
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2013-06-17 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Comparison of the measures of ovarian reserve (AMH, FSH and E2) to that of health controls | Up to 12 months
  Compared using the Wilcoxon rank-sum test or the two sample t-test after appropriate transformation. Analysis of covariance will be used to adjust these comparisons for covariates including age, race, dose of alkylating agent and use of hormone medications.
Degree of change in AMH, FSH, and E2 defined as the ratio of baseline minus end of therapy (EOT) measurement over baseline | Baseline up to end of chemotherapy
  Evaluated using Wilcoxon signed rank test or a paired t-test after appropriate normalizing transformation.
Degree of recovery of AMH, FSH, and E2 in the post-therapy phase | Up to 12 months
  Generalized estimating equation (GEE) will be used to model the change as a function of time.

SECONDARY OUTCOMES:
Rate of AOF | Up to 12 months
  Describe the number of patients with AOF as measured at 12 months by an FSH > 40 divided by the total population.
Collect blood samples for future evaluation of drug metabolizing Describe number of samples enzyme polymorphisms | At enrollment (or diagnosis) and Day 5 post enrollment
  Describe the number of samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Levine, Principal Investigator — Children's Oncology Group
Locations (107):
- United States (97):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (10):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec